CLINICAL TRIAL: NCT05834400
Title: Lymphatic System Stimulation and Fluid Overload Symptoms in Patients With Heart Failure
Brief Title: Lymphatic System Stimulation in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Rida Gharzeddine, PhD, RN, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro2022001875
Record Dates: First submitted 2023-04-03; First posted 2023-04-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac Edema; Self-care; Exercise Movement Techniques
MeSH Terms: conditions — Heart Failure; Edema, Cardiac

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Optimal Lymph Flow (TOLF) (Experimental): Participants in this arm perform lymphatic exercise training AND daily monitoring of fluid overload symptoms for 4 weeks
  Interventions: Behavioral: The Optimal Lymph FLow (TOLF); Behavioral: Daily Monitoring
- Daily Monitoring (Active Comparator): Participants in this arm will only perform daily monitoring of fluid overload symptoms including weight, heart rate, and blood pressure for 4 weeks. Participants will NOT perform TOLF in this arm.
  Interventions: Behavioral: Daily Monitoring

INTERVENTIONS:
Behavioral: The Optimal Lymph FLow (TOLF) — Participants in TOLF intervention will complete initial in-person 40-minute session on TOLF lymphatic exercise training and daily monitoring, and 3 virtual 15-minute telehealth sessions to enhance their skills over the course of 4 weeks. These sessions will be conducted by the TOLF interventionist of the study. For 4-week study duration, participants will be asked to practice the set of 8 lymphatic exercises twice a day.
  Arms: The Optimal Lymph Flow (TOLF)
Behavioral: Daily Monitoring — Participants will complete initial in-person training on daily monitoring of weight, heart rate and blood pressure, fluid overload symptoms; and 3 conferencing coaching sessions conducted by the monitoring coach to enhance their skills. Over the course of 4 weeks, Participants will monitor these daily fluid overload parameters and symptoms

SUMMARY:
The goal of this pilot clinical trial is to obtain preliminary data on the effects of lymphatic exercise training in patients with heart failure. The main question[s] it aims to answer are:

1. Does performing lymphatic exercise decrease fluid overload symptoms (shortness of breath, lower legs swelling, fatigue), thoracic fluid content, and body fluid level?
2. Does performing lymphatic exercise improve sleep and quality of life (QOL)?

Participants with heart failure will be randomly assigned into two groups:

Group 1 will receive training on lymphatic exercises, and will perform these training for 4 weeks. This group will also be trained to monitor daily their weight, heart rate and blood pressure, and fluid overload symptoms.

Group 2 will be trained to daily monitor their weight, heart rate and blood pressure, and fluid overload symptoms. This group will not perform the lymphatic exercises.

Researchers will compare the two groups at the baseline and after delivering the 4 week-interventions to see

1. if lymphatic exercise helped decrease symptoms associated with fluid overload like shortness of breath, lower leg swelling, and fatigue.
2. if lymphatic exercises decreased thoracic fluid content and total body fluid level .
3. if the lymphatic exercise helped improve sleep and quality of life (QOL).

DETAILED DESCRIPTION:
Heart failure (HF) is a growing public health problem affecting 6.2 million people in the United States. Fluid overload, the hallmark of HF, refers to a progressive body fluid retention or redistribution that impedes multiple body system functions and leads to symptoms of pulmonary congestion (e.g., dyspnea, orthopnea, coughing, or wheezing) and systemic venous congestion (e.g., edema, fatigue, bodily pain, and gastrointestinal disturbance). Fluid overload symptoms are highly prevalent and burdensome, profoundly limiting patients' daily functioning and well-being. The occurrence or exacerbation of fluid overload symptoms is the major reason for patients with HF to be admitted or readmitted to hospital and causes patients' distress and poor QOL, imposing considerable burdens on the individual, family, and health care system.

The surveillance and management of worsening fluid overload symptoms is the cornerstone of HF care. Recent research on the role of lymphatic system in the pathogenesis of cardiovascular diseases has highlighted new therapeutic perspectives of fluid volume removal or fluid overload management in HF. If fluid is not drained at the same rate as it leaks, the painful and debilitating condition of fluid overload would develop. Prior work on lymphedema and symptoms related to lymph fluid accumulation in breast cancer patients showed efficacy in reduction of swelling, lymph fluid accumulation, reversed mild lymphedema, and improvement in pain severity, swelling severity, psychological distress, and QOL in these women. A recently published systematic review and meta-analysis summarizes data from 17 RCTs covering 1086 participants and demonstrated that peripheral muscle contracted exercises (e.g., aerobic exercises) can help to reduce the fluid overload symptom of dyspnea and edema. Thus, exercises focusing on optimizing lymph flow is a potential therapeutic approach to management of fluid overload symptoms in HF.

The specific aims of this study are to:

Aim1: Assess the feasibility and acceptability of lymphatic exercise training and obtaining data on fluid overload symptoms and body fluid level in adult patients with HF over training sessions. Feasibility will be assessed via (a) study accrual, (b) protocol adherence, and (c) retention.

Aim 2: Provide preliminary data for estimation of the effects of lymphatic exercise training on fluid overload symptoms and body fluid level at post-training compared to daily monitoring group.

Aim 3: Explore the effects of lymphatic exercise training on sleep, quality of life (QOL), and he number of abnormal weight fluctuations, at post-training compared to daily monitoring group.

Research Design and Methods Design. We will use a prospective Randomized Controlled Trial (RCT) design to assess the feasibility, acceptability, and outcome patterns suggesting efficacy of a TOLF Lymphatic Exercise Training for Fluid Overload Symptom Management protocol. This study will be conducted at the Cooper University Health Care (Cooper) with 80 adult HF patients.

Study Population. Patients aged 18 to 80 years, hospitalized due to fluid overload with a primary diagnosis of HF in the chronic or stable phase.

Research Procedures A total of 80 participants will be recruited. Following consent and baseline assessment, 80 participants will be randomly assigned in equal allocation to one of two conditions: 1) TOLF + Daily Monitoring (DM) or 2) DM. Our research evaluator will not be involved in recruitment or have other contact with participants; they will be blinded to participant randomization and conduct all study procedures where blinding is indicated (e.g., assessments). Additionally, all efforts will be made for study staff and participants to be blinded to participant condition.

Recruitment and Informed Consent. All recruitment procedures will comply with HIPAA guidelines. The recruitment procedure will be as follows: Potential participants will be identified through electronic medical record review or their medical team. Once a potential participant has been identified, their primary physician will be contacted for permission to attempt to recruit the participant for this study. If the physician agrees, potential participants will be told about the study by a member of the medical staff and asked if they would be willing to talk with a member of the study team. Once a potential subject agrees, a member of the study team at Cooper will approach the patient. At this time, the member of the study team will describe the study in detail, provide the patient with consent forms, and offer to answer any questions about the study. Once a patient has consented, they will complete the first study assessment before he/she discharged from the hospital to home.

RCT Randomization. Following consent and baseline assessment, 80 participants will be randomly assigned in equal allocation to one of two conditions: 1) TOLF + Daily Monitoring (DM) or 2) DM. Randomization will be blocked by NYHA functional class II, III, IV and gender to ensure reasonable balance in each treatment condition. The data programmer on this study who is not involved with recruitment will randomly draw a number of 1 or 2 to be given the participant's study number (not name) to randomize the participant. Our research evaluator will not be involved in recruitment or have other contact with participants; they will be blinded to participant randomization and conduct all study procedures where blinding is indicated (e.g., assessments). Additionally, all efforts will be made for study staff and nurses and physicians to be blinded to participant condition. Participants who do not have a smartphone will be loaned a cellular phone with Internet access to the mHealth features: video-conferencing, fluid overload symptom management skill content, TOLF lymphatic exercise videos.

Treatment Conditions. It is expected that participants either in TOLF+DM or DM groups will complete initial in-person 40-minute session, and 3 virtual 15-minute telehealth video-sessions over the course of 4 weeks.

Daily Monitoring (DM): Participants will complete initial in-person training on daily monitoring of weight, heart rate and blood pressure, fluid overload symptoms; and 3 video-conferencing coaching sessions conducted by the monitoring coach to enhance their skills.

The-Optimal-Lymph-Flow (TOLF): Patients in TOLF intervention will complete initial in-person 40-minute session on TOLF lymphatic exercise training and daily monitoring, and 3 virtual 15-minute telehealth video-sessions to enhance their skills over the course of 4 weeks. These sessions will be conducted by the TOLF interventionist of the study. For 4-week study duration, participants will be asked to practice the set of 8 lymphatic exercises twice a day.

Therapist Training. TOLF and DM skills training sessions will be delivered by nurses with experience working with HF patients. Treatment strategies will be taught through didactic instruction, audio-/video-recorded illustration of techniques, and role-play.

Procedures to Ensure Consistency of TOLF Treatment. To ensure consistency with the intervention protocol: 1) therapist will follow a treatment manual, 2) weekly supervision will occur, 3) sessions will be audio-recorded and reviewed during supervision and feedback provided, and 4) ratings of treatment adherence and competence will be conducted.

Timing and Frequency of data collection:

Demographics and baseline data will be collected in Cooper University Health Care (Cooper) Cardiac Unit before patients are discharged. Participants will be asked for a research visit to Cooper University Health Care (Cooper) on week 5 to collect post intervention data.

During the intervention duration, participants will be asked to text their weight, heart rate and blood pressure daily, and keep a daily log that will bring with them on week 5 Research Staff Training Research evaluator. The research evaluator will be a recruited nurse who will collect self-reported and objective data from participants. Research evaluator/ data collector will be trained on how to ask and explain questions in the questionnaires, and how to use objective devices to collect objective data on fluid content and level. Training will include didactic instruction, audio-/video-recorded illustration of techniques, and role-play Therapist Training. TOLF and DM skills training sessions will be delivered by two research assistant nurses who had experience working with HF patients. One therapist will be the interventionist and the second will be the monitoring coach to avoid contamination. Treatment strategies will be taught through didactic instruction, audio-/video-recorded illustration of techniques, and role-play.

Procedures to Ensure Consistency of TOLF Treatment. To ensure consistency with the intervention protocol: 1) therapist will follow a treatment manual, 2) weekly supervision will occur, 3) sessions will be audio-recorded and reviewed during supervision and feedback provided, and 4) ratings of treatment adherence and competence will be conducted.

Data Analysis Aim 1 Analyses. Feasibility will be assessed by examining accrual, adherence, and attrition. Accrual will be indicated by meeting the recruitment goal of 80 participants in 24 months. Descriptive statistics will be reported on the number of HF patients screened and determine rates of non-eligibility and refusal. Adherence will be indicated by calculating the proportion successfully completing all intervention sessions within the TOLF+DM arm and the proportion completing post-treatment assessments within each arm. 80% completed intervention sessions and 80% completed assessments will serve as our feasibility benchmark. With a sample size of 50, we will be able to estimate a rate of 80% to within the 95% confidence interval width of +/- 11%. So, if less than 69% of participants complete all intervention sessions and assessments, TOLF+DM will not be considered feasible. Attrition will be indicated by 80% of consented participants completing the study protocol (i.e., remain enrolled). Acceptability will be indicated by 80% of patients reporting satisfaction with TOLF+DM (Mean=7) on the CSQ. Aim 2 & 3 Analyses. Between-group effect sizes will be used to evaluate treatment effects on fluid overload symptoms, TFCI, body fluid level, hospital readmission, the number of abnormal weight fluctuations, and QOL. Between-group effect sizes will provide an index of relative change for TOLF+DM participants vs. DM participants. Because small samples can differ on pretest scores, effect sizes will be calculated by first creating change scores for each person. The between-group effect size will then be calculated by subtracting the average DM group change score from the average TOLD+DM change score, and dividing this difference by the standard deviation of the pooled treatment/control group's change score. This study is not designed to make conclusions about efficacy without further study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HF with New York Heart Association (NYHA) functional class II, III, or IV
* Willing and able to complete the home-based TOLF program upon discharge from the hospital to home

Exclusion Criteria:

* Severe liver or kidney insufficiency or malignant tumors
* A terminal condition with a life expectancy of < 6 months
* Received or waiting for heart transplantation
* Pregnancy
* Cognitive impairment (e.g., dementia)
* Severe psychiatric condition (psychotic disorder, severe depression, suicidal intent)
* Inability to converse in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Fluid Overload Symptoms | 4 weeks
  Fluid overload symptoms include shortness of breath, difficulty breathing when lying flat, cough, lack of energy, swelling of legs or ankles, and waking up breathless at nigh swelling of the lower extremities. These symptoms are measured by The Memorial Symptom Assessment Scale - Heart Failure (MSAS-HF). Individual scores are summed for each symptom present, rating frequency, severity, and distress to obtain a total symptom score for each symptom with a possible range of 0-13. Higher scores indicate greater symptom burden.
Thoracic Fluid Content | 4 weeks
  Will be assessed by the FDA approved, non-invasive remote dielectric sensing (ReDS) (Sensible Medical Innovations, Ltd, Israel). ReDS uses low-power electromagnetic signals emitted between 2 sensors (1 each on the anterior and posterior body surfaces) embedded in a wearable vest
Body Fluid Content | 4 weeks
  Will be measured by stand-on bioimpedance analysis (BIA) device (InBody 570, Biospace Co., Ltd., Cerritos, CA, USA). Intracellular and extracellular fluid levels are measured to determine total body fluid levels. These measures will be combined to determine the ratio of extracellular fluid to the total body fluid to indicate whether body fluids are balanced. Normal ratios range from 0.36 to 0.39, and higher ratios are indicative of fluid retention and edema.

SECONDARY OUTCOMES:
Health related Quality of Life | 4 weeks
  Will be measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The Minnesota Living with Heart Failure Questionnaire (MLHFQ) provides a total score (range 0-105), with higher scores indicating worse quality of life
Sleep Quality | 4 weeks
  Sleep quality is measured with the Pittsburgh Sleep Quality Index (PSQI). The scores are summed to yield a total score ranging from 0 to 21, with the higher total score (referred to as global score) indicating worse sleep quality.
Insomnia Severity | 4 weeks
  Insomnia severity is measured by Insomnia Severity Index (ISI). Total score ranges from 0-28 with higher scores indicating worse insomnia severity.
Daytime sleepiness | 4 weeks
  Daytime sleepiness is measured by The Epworth Sleepiness Scale (ESS) where the total score ranges from 0-24. Scores of 11-24 represent increasing levels of 'excessive daytime sleepiness.

OTHER OUTCOMES:
Number of abnormal weight fluctuations | 4 weeks
  Will be measured by daily logs reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Rida Gharzeddine, PhD, Principal Investigator — Rutgers, The State University of New Jersery
Locations (1):
- Cooper University Health Care (Cooper), Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu MR, Li Y, Conway C, Masone A, Fang J, Lee C. The Effects of Exercise-Based Interventions on Fluid Overload Symptoms in Patients with Heart Failure: A Systematic Review and Meta-Analysis. Biomedicines. 2022 May 11;10(5):1111. doi: 10.3390/biomedicines10051111. PMID 35625848
- [Background] Liu F, Li F, Fu MR, Zhao Q, Wang Y, Pang D, Yang P, Jin S, Lu Q. Self-management Strategies for Risk Reduction of Subclinical and Mild Stage of Breast Cancer-Related Lymphedema: A Longitudinal, Quasi-experimental Study. Cancer Nurs. 2021 Nov-Dec 01;44(6):E493-E502. doi: 10.1097/NCC.0000000000000919. PMID 34694088
- [Background] Fu MR, Axelrod D, Guth AA, Scagliola J, Rampertaap K, El-Shammaa N, Qiu JM, McTernan ML, Frye L, Park CS, Yu G, Tilley C, Wang Y. A Web- and Mobile-Based Intervention for Women Treated for Breast Cancer to Manage Chronic Pain and Symptoms Related to Lymphedema: Results of a Randomized Clinical Trial. JMIR Cancer. 2022 Jan 17;8(1):e29485. doi: 10.2196/29485. PMID 35037883